CLINICAL TRIAL: NCT02129777
Title: A Multi-Centre, Randomized, Double-Blind, Placebo-Controlled, Dose-Finding and Proof of Concept Study, to Assess the Efficacy, Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of Namilumab/MT203 at 4 Different Subcutaneous Doses - Together With an Open-Label, Dose-Escalated Extension to Assess Safety and Efficacy of One Year Treatment - in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Efficacy and Safety of Namilumab (MT203) for Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M1-1188_203; U1111-1146-1219 (Other: WHO); 2013-002806-30 (EudraCT Number); 172235 (Registry Identifier: HC-CTD)
Record Dates: First submitted 2014-04-14; First posted 2014-05-02 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-02

CONDITIONS: Plaque Psoriasis
Keywords: Drug therapy
MeSH Terms: interventions — namilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Blinded period: Namilumab 300 mg + namilumab 150 mg (Experimental): Namilumab 300 mg (2 separate injections of 150 mg), subcutaneous injection, on Day 1, followed by namilumab 150 mg subcutaneous injection, on Days 15, 43 and 71.
  Interventions: Drug: Namilumab
- Blinded period: Namilumab 160 mg + namilumab 80 mg (Experimental): Namilumab 160 mg (2 separate injections of 80 mg), subcutaneous injection, on Day 1, followed by namilumab 80 mg subcutaneous injection, on Days 15, 43 and 71.
  Interventions: Drug: Namilumab
- Blinded period: Namilumab 100 mg + namilumab 50 mg (Experimental): Namilumab 100 mg (2 separate injections of 50 mg), subcutaneous injection, on Day 1, followed by namilumab 50 mg subcutaneous injection, on Days 15, 43 and 71.
  Interventions: Drug: Namilumab
- Blinded period: Namilumab 40 mg + namilumab 20 mg (Experimental): Namilumab 40 mg (2 separate injections of 20 mg), subcutaneous injection, on Day 1, followed by namilumab 20 mg subcutaneous injection, on Days 15, 43 and 71.
  Interventions: Drug: Namilumab
- Blinded period: Placebo (Placebo Comparator): Placebo (2 separate injections), subcutaneous injection, on Day 1, followed by placebo, subcutaneous injection, on Days 15, 43 and 71.
  Interventions: Drug: Placebo
- Open label: Namilumab 80 mg (Experimental): Namilumab 80 mg subcutaneous injection, at Week 0 and every 4 weeks thereafter up to 52 weeks (active extension period) - if appropriate on the basis of treatment response.
  Interventions: Drug: Namilumab
- Open label: Namilumab 150 mg (Experimental): Namilumab 150 mg, subcutaneous injection, from Week 8 and then every 4 weeks thereafter up to 52 weeks (active extension period) - if appropriate on the basis of treatment response.
  Interventions: Drug: Namilumab

INTERVENTIONS:
Drug: Namilumab — Namilumab subcutaneous injection
  Other Names: MT203
  Arms: Blinded period: Namilumab 100 mg + namilumab 50 mg; Blinded period: Namilumab 160 mg + namilumab 80 mg; Blinded period: Namilumab 300 mg + namilumab 150 mg; Blinded period: Namilumab 40 mg + namilumab 20 mg; Open label: Namilumab 150 mg; Open label: Namilumab 80 mg
Drug: Placebo — Placebo subcutaneous injection
  Arms: Blinded period: Placebo

SUMMARY:
The purpose of this study is to establish proof of efficacy for namilumab in moderate to severe plaque psoriasis, measured as Psoriasis Area and Severity Index (PASI)75 response rate at Week 12.

DETAILED DESCRIPTION:
The drug tested in this study is called namilumab. Namilumab was tested to prove its effectiveness in treating moderate to severe chronic plaque psoriasis. This study looked at improvement of plaque psoriasis in participants who take namilumab.

The study enrolled 122 participants. Participants were randomly assigned (by chance, like flipping a coin) to one of five treatment groups that were undisclosed to the patient and study doctor during the study (unless there was an urgent medical need):

* Namilumab subcutaneous injection 300 mg Day 1, 150 mg Days 15, 43 and 71
* Namilumab subcutaneous injection 160 mg Day 1, 80 mg Days 15, 43 and 71
* Namilumab subcutaneous injection 100 mg Day 1, 50 mg Days 15, 43 and 71
* Namilumab subcutaneous injection 40 mg Day 1, 20 mg Days 15, 43 and 71
* Placebo (dummy inactive subcutaneous injection) - this is a liquid solution that looks like the study drug but has no active ingredient Days 1, 15, 43 and 71.

This study consisted of two parts. Eligible participants received 10 weeks of treatment with double-blinded study medication, followed by an extended treatment period (active extension period, intended to be 52 weeks) with open-label study medication. At Week 12, participants were assessed for primary endpoint response, which determined the course of their progression through the open-label treatment period. Participants who showed >=75% reduction of Baseline (Day 1) PASI at Week 12, "Responders", began a washout interval (for a maximum of 24 weeks) with no use of study medication: this interval continued until a partial (25%) loss of Week 12 treatment response is recorded in assessments conducted on a 2-weekly basis - thereby prompting the start of dosing with open-label (OL) study medication (Day 0 OL through Week 52 OL). In contrast, participants who did not show >=75% reduction of Baseline PASI score at Week 12, "Partial/Non-Responders", began the open-label extension period 4 weeks after the final dose of blinded study medication.

Participants were then followed-up through an 18-week post-treatment assessment period during which no medication was given. During the open-label extension period participants began dosing with 80 mg namilumab; however, if an inadequate treatment response was recorded, then dose escalation to 150 mg namilumab was implemented.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female aged 18 to 70 years, inclusive.
2. Is suffering from active but clinically stable plaque psoriasis (for at least 6 months) involving >=10% of their body surface area and Psoriasis Area and Severity Index (PASI) score >=12.
3. Must have been a candidate for, or have received, >= phototherapy or systemic psoriasis therapy.
4. A male participant who is non-sterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of the informed consent throughout the duration of the study (including the treatment period and 18 weeks after last dose of study medication).
5. A female participant of childbearing potential who is sexually active with a non-sterilized male partner agrees to routinely use adequate contraception from signing of the informed consent throughout the duration of the study (including the treatment period and 18 weeks after last dose of study medication).
6. In the opinion of the investigator, is capable of understanding and complying with protocol requirements.
7. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written informed consent form and any required privacy authorization prior to the initiation of any study procedures.

Exclusion Criteria:

1. Has received any investigational agent during an interval equivalent to 5 half- lives for that agent agent - or an interval of 30 days if longer - prior to the study Baseline clinic visit, or is participating / plans to participate in any other clinical trial during this study.
2. Has received namilumab, any other Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) / GM-CSF receptor or granulocyte stimulating factor (G-GSF) signaling inhibitor either in a previous clinical study or as a therapeutic agent.
3. Is required to take excluded medications.
4. Has a history of hypersensitivity or allergies to namilumab or any of the contents of the formulation.
5. Has other forms of psoriasis (eg drug-induced psoriasis, pustular, erythrodermic, exfoliative, inverse and/or guttate psoriasis).
6. Evidence of skin conditions other than psoriasis (eg, eczema) at the time of the Screening clinic visit, or between the Screening visit and study drug initiation, that would interfere with evaluations of the effect of investigational product on psoriasis.
7. Has a history or evidence of a clinically significant disorder (including but not limited to cardiopulmonary, oncologic, renal, metabolic, hematologic or psychiatric), condition or disease that, in the opinion of the investigator and Takeda physician would pose a risk to participant safety or interfere with the study evaluation, procedures or completion.
8. Evidence of clinically uncontrolled respiratory disease (including sarcoidosis) on the basis of data from the subjects' respiratory assessments - including chest X-ray, lung function tests (forced expiratory volume in one second [FEV1], forced vital capacity [FVC], peak expiratory flow rate [PEFR]) and pulse oximetry performed at Screening. The subjects must have saturation of peripheral oxygen (SpO2) ≥ 94%, FEV1 and/or FVC ≥ 60 % of predicted values at Screening and Baseline and no uncontrolled lung disease. Subject treatment initiated or modified to control lung disease within 24 weeks prior to Screening must be considered exclusionary.
9. History of clinically significant interstitial lung disease - e.g. chronic or recurrent pulmonary infection where macrophages are important for the clearance of the infection (such as Pneumocystis (carinii) jiroveci pneumonia, allergic bronchopulmonary aspergillosis, Nocardia infections, Actinomyces infection).
10. Presence or history of active tuberculosis (TB) or latent TB infection, where no anti-TB treatment has been given or where successful completion of an appropriate course of anti-TB therapy cannot be documented.
11. A positive QuantiFERON-TB Gold test and / or evidence of active or latent TB by chest X- ray, not accompanied by initiation of an approved regimen of anti-TB therapy at least 12 months prior to the Baseline clinic visit.
12. Has a history of severe chronic obstructive pulmonary disease (COPD) and / or history of severe COPD exacerbation(s), or a history of asthma with exacerbations requiring hospitalization, within the last 12 months prior to the Screening visit.
13. History of methotrexate treatment-associated lung toxicity.
14. Has a history of cancer within the last 10 years except for adequately managed basal cell or squamous cell carcinoma of the skin or in situ carcinoma of the cervix treated and considered cured.
15. Has a history of treatment with anti-cancer chemotherapy (e.g. alkylating agents, anti-metabolites, purine analogues) and/or monoclonal antibodies, or has received GM-CSF / G-CSF treatment associated with chemotherapy within the last 5 years.
16. Has an underlying condition that predisposes to infections (eg immunodeficiency, history of poorly controlled diabetes, splenectomy).
17. Has any clinically significant illness within 4 weeks prior to the first dose of study medication or during the study - including acute or chronic infectious disease, which may influence the outcome of the study.
18. Has a known history of infection with hepatitis B virus, hepatitis C virus, or human immunodeficiency virus (HIV), or has serological findings at the Screening visit which indicate active or latent hepatitis B, hepatitis C or HIV infection.
19. Has, in the judgment of the investigator, clinically significant abnormal clinical laboratory parameters at Screening including, but not limited to: Hemoglobin <8.5 g/dL, Neutrophils <1500/mm^3, Platelet count <75 000 cells/mm^3 and AST or ALT >2 x ULN.
20. Has a history of drug abuse (defined as any illicit drug use), or a history of alcohol abuse within 2 years prior to the Screening visit.
21. Any other condition that, in the judgment of the investigator, might cause this study to be detrimental to the participant's health.
22. If female, is (a) pregnant / lactating / intending to become pregnant before or within the period of 18 weeks immediately after receiving the last dose of study medication; (b) intending to donate ova during this time period.
23. Intends to donate sperm during the course of this study or within a period of 18 weeks after receiving the last dose of study medication.
24. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee involved in conduct of this study (eg, spouse, parent, child, sibling), or may consent under duress.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Clinical Science, Study Director — Takeda
Locations (10):
- Canada (10):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Barrie, Ontario
  - Hamilton, Ontario
  - Markham, Ontario
  - North Bay, Ontario
  - Peterborough, Ontario
  - Richmond Hill, Ontario
  - Waterloo, Ontario
  - Québec, Quebec

REFERENCES:
- [Derived] Papp KA, Gooderham M, Jenkins R, Vender R, Szepietowski JC, Wagner T, Hunt B, Souberbielle B; NEPTUNE investigators. Granulocyte-macrophage colony-stimulating factor (GM-CSF) as a therapeutic target in psoriasis: randomized, controlled investigation using namilumab, a specific human anti-GM-CSF monoclonal antibody. Br J Dermatol. 2019 Jun;180(6):1352-1360. doi: 10.1111/bjd.17195. Epub 2018 Nov 2. PMID 30207587

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled into the double-blind treatment evaluation at 17 investigative sites in Canada, Denmark, Germany, Latvia, and Poland. Only those sites in Denmark, Latvia and Poland participated in the extension period which included open-label treatment with study medication.
Pre-assignment Details: Participants with diagnosis of moderate to severe plaque psoriasis without clinically significant lung/respiratory disorders were screened for enrollment into the study.To fulfill screening requirements,chest X-ray was carried out prior to Baseline visit which included assignment to the double-blind study treatment and first dosing with study drug.
Groups:
- Double-Blind Period: Placebo: Namilumab-matching placebo solution (2 separate injections) subcutaneously on Day 1, followed by namilumab-matching placebo, single injection, subcutaneously at Weeks 2, 6 and 10 during the double-blind period.
- Double-Blind Period: Namilumab 20 mg: Namilumab 40 milligram (mg) injection (2 separate injections of 20 mg) subcutaneously on Day 1, followed by namilumab 20 mg, single injection, subcutaneously at Weeks 2, 6 and 10 during the double-blind period.
- Double-Blind Period: Namilumab 50 mg: Namilumab 100 mg injection (2 separate injections of 50 mg) subcutaneously on Day 1, followed by namilumab 50 mg, single injection, subcutaneously at Weeks 2, 6 and 10 during the double-blind period.
- Double-Blind Period: Namilumab 80 mg: Namilumab 160 mg injection (2 separate injections of 80 mg) subcutaneously on Day 1, followed by namilumab 80 mg, single injection, subcutaneously at Weeks 2, 6 and 10 during the double-blind period.
- Double-Blind Period: Namilumab 150 mg: Namilumab 300 mg injection (2 separate injections of 150 mg) subcutaneously on Day 1, followed by namilumab 150 mg, single injection, subcutaneously at Weeks 2, 6 and 10 during the double-blind period.
- Open-Label Period: Namilumab 80 mg: Namilumab 80 mg, single injection, subcutaneously, every 4 weeks for 52 weeks during the open-label period on the basis of treatment response.
- Open-Label Period: Namilumab 150 mg: Namilumab 150 mg, single injection, subcutaneously from Week 8 and then every 4 weeks for 52 weeks during the open-label period on the basis of treatment response.
Period: Double-Blind Period
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg | Open-Label Period: Namilumab 80 mg | Open-Label Period: Namilumab 150 mg
Started | 24 | 24 | 24 | 25 | 25 | 0 | 0
Completed | 17 | 16 | 20 | 18 | 18 | 0 | 0
Not Completed | 7 | 8 | 4 | 7 | 7 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 3 | 2 | 3 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 3 | 1 | 0 | 3 | 2 | 0 | 0
Not completed — Other | 1 | 2 | 0 | 0 | 0 | 0 | 0
Period: Open-Label Period
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg | Open-Label Period: Namilumab 80 mg | Open-Label Period: Namilumab 150 mg
Started | 0 | 0 | 0 | 0 | 0 | 12 | 48
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 12 | 48
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 3
Not completed — Study Termination | 0 | 0 | 0 | 0 | 0 | 10 | 39

BASELINE CHARACTERISTICS:
Population: Randomized set included all participants randomized in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg | Total
Number analyzed (Participants) | 24 | 24 | 24 | 25 | 25 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (15.20) | 41.1 (11.28) | 42.3 (10.92) | 39.0 (12.04) | 39.8 (9.62) | 40.6 (11.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 5 | 7 | 13 | 38
  Male | 15 | 20 | 19 | 18 | 12 | 84
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic or Latino | 10 | 10 | 12 | 12 | 12 | 56
  Unknown or Not Reported | 14 | 14 | 12 | 13 | 13 | 66
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2 | 1 | 2 | 2 | 4 | 11
  Black or African American | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 1
  White | 22 | 22 | 21 | 23 | 21 | 109
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 10 | 12 | 12 | 12 | 56
  Denmark | 0 | 1 | 0 | 0 | 1 | 2
  Germany | 0 | 0 | 0 | 0 | 1 | 1
  Latvia | 5 | 5 | 2 | 3 | 2 | 17
  Poland | 9 | 8 | 10 | 10 | 9 | 46
Height [Mean (Standard Deviation); unit: centimeter] | 172.3 (10.83) | 176.1 (7.73) | 176.5 (7.81) | 176.8 (8.59) | 168.1 (10.28) | 173.9 (9.61)
Weight [Mean (Standard Deviation); unit: kilogram] | 87.46 (22.864) | 88.26 (22.033) | 97.84 (33.643) | 95.50 (25.056) | 82.32 (24.634) | 90.25 (26.156)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 29.16 (6.112) | 28.25 (5.936) | 31.26 (9.532) | 30.53 (7.641) | 29.01 (8.093) | 29.64 (7.539)
Smoking Classification [Number; unit: participants]
  Never Smoked | 7 | 11 | 9 | 13 | 12 | 52
  Current Smoker | 8 | 5 | 9 | 7 | 5 | 34
  Ex-Smoker | 9 | 8 | 6 | 5 | 8 | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving 75 Percent Reduction From Baseline Psoriasis Area and Severity Index (PASI) Score (PASI75 Response) at Week 12
Description: PASI is an assessment of psoriasis lesion severity and affected body area combined into single score. The body was divided into 4 sections: head (h), trunk (t), upper (u) and lower (l) extremities. For each section, percent body surface area (A) involved was estimated: 0= No involvement to 6= 90-100 percent (%). Severity was estimated by clinical signs: erythema (E), induration (I), and desquamation (D); scale: 0= no symptoms to 4= very marked. Final PASI = 0.1(Eh + Ih + Dh)Ah + 0.3(Et + It + Dt)At + 0.2(Eu + Iu + Du)Au + 0.4(El + Il + Dl)Al where head: 0.1, upper extremities (arms): 0.2, trunk: 0.3, lower extremities (legs): 0.4 (corresponding to approximately 10%, 20%, 30%, and 40% of body surface area, respectively); total possible score range: 0= no disease to 72= maximal disease. Participants showing at least 75% reduction in PASI score relative to baseline PASI Score are reported.
Time Frame: Week 12
Population: Full analysis set (FAS) where baseline and Week 12 assessment were available. FAS included all randomized and treated participants who had at least one valid post-baseline assessment of PASI in the double-blind period.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg
Number analyzed (Participants) | 23 | 21 | 22 | 19 | 20
percentage of participants | 8.7 | 9.5 | 0 | 5.3 | 0
Statistical Analysis 1: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 20 mg; Cochran-Mantel-Haenszel (CMH) P-values are from a CMH Chi-Square test using a 2*2 contingency table of treatment and responder status controlling for visit; Test type: Superiority or Other; p = 0.925, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.008, 95% CI 2-sided [-0.162 to 0.179] — Risk difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 2: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 50 mg; CMH P-values are from a CMH Chi-Square test using a 2*2 contingency table of treatment and responder status controlling for visit; Test type: Superiority or Other; p = 0.162, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.087, 95% CI 2-sided [-0.202 to 0.028] — Risk difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 3: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 80 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.671, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.034, 95% CI 2-sided [-0.187 to 0.118] — Risk difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 4: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 150 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.182, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.087, 95% CI 2-sided [-0.202 to 0.028] — Risk difference (namilumab - placebo) and corresponding 95% confidence interval were reported

2. Secondary Outcome: Percentage of Participants Achieving 75 Percent Reduction From Baseline PASI Score (PASI75 Response) at Weeks 2, 4, 6, and 10
Description: as for outcome 1
Time Frame: Weeks 2, 4, 6 and 10
Population: FAS where baseline and specified post-baseline assessment were available. FAS included all randomized and treated participants who had at least one valid post-baseline assessment of PASI in the double-blind period.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg
Number analyzed (Participants) | 24 | 24 | 24 | 25 | 25
percentage of participants
  Week 2 (n= 24, 24, 24, 25, 25) | 0 | 0 | 0 | 0 | 0
  Week 4 (n= 24, 24, 23, 24, 24) | 0 | 0 | 4.3 | 0 | 0
  Week 6 (n= 23, 23, 24, 24, 23) | 4.3 | 8.7 | 4.2 | 4.2 | 0
  Week 10 (n= 22, 22, 24, 24, 22) | 9.1 | 4.5 | 0 | 4.2 | 0

3. Secondary Outcome: Change From Baseline in PASI Score at Weeks 2, 4, 6, 10, and 12
Description: PASI is an assessment of psoriasis lesion severity and affected body area combined into single score. The body was divided into 4 sections: head (h), trunk (t), upper (u) and lower (l) extremities. For each section, percent body surface area (A) involved was estimated: 0= No involvement to 6= 90-100 percent (%). Severity was estimated by clinical signs: erythema (E), induration (I), and desquamation (D); scale: 0= no symptoms to 4= very marked. Final PASI = 0.1(Eh + Ih + Dh)Ah + 0.3(Et + It + Dt)At + 0.2(Eu + Iu + Du)Au + 0.4(El + Il + Dl)Al where head: 0.1, upper extremities (arms): 0.2, trunk: 0.3, lower extremities (legs): 0.4 (corresponding to approximately 10%, 20%, 30%, and 40% of body surface area, respectively); total possible score range: 0= no disease to 72= maximal disease.
Time Frame: Baseline, Weeks 2, 4, 6, 10, and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg
Number analyzed (Participants) | 24 | 24 | 24 | 25 | 25
units on a scale
  Baseline (n=24, 24, 24, 25, 25) | 18.6 (1.65) | 19.1 (1.57) | 20.9 (1.62) | 17.4 (1.57) | 17.3 (1.52)
  Change at Week 2 (n=24, 24, 24, 25, 25) | -2.2 (0.70) | -1.7 (0.67) | -1.2 (0.69) | -2.1 (0.67) | -1.4 (0.65)
  Change at Week 4 (n=24, 24, 23, 24, 24) | -3.6 (0.92) | -2.8 (0.90) | -1.9 (0.92) | -2.4 (0.90) | -2.2 (0.89)
  Change at Week 6 (n=23, 23, 24, 24, 23) | -5.1 (1.13) | -3.6 (1.10) | -1.4 (1.11) | -2.4 (1.10) | -2.4 (1.10)
  Change at Week 10 (n=22, 22, 24, 24, 22) | -6.4 (1.30) | -4.6 (1.29) | -3.2 (1.28) | -3.2 (1.27) | -3.0 (1.28)
  Change at Week 12 (n=23, 21, 22, 19, 20) | -6.3 (1.27) | -4.9 (1.26) | -4.4 (1.25) | -3.3 (1.26) | -3.4 (1.26)
Statistical Analysis 1: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 20 mg; Week 12: Post-baseline least squares means and p-values were from a MMRM model with main effect of study site, treatment, visit and interaction between visit and treatment as fixed effects, baseline value as a covariate with an unstructured covariance structure; Test type: Superiority or Other; p = 0.435, MMRM; LS Mean Difference = 1.4, 95% CI 2-sided [-2.1 to 4.9], Standard Error of Mean 1.75 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 2: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 50 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.279, MMRM; LS Mean Difference = 1.9, 95% CI 2-sided [-1.6 to 5.4], Standard Error of Mean 1.74 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 3: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 80 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.085, MMRM; LS Mean Difference = 3.0, 95% CI 2-sided [-0.4 to 6.5], Standard Error of Mean 1.74 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 4: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 150 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.110, MMRM; LS Mean Difference = 2.8, 95% CI 2-sided [-0.7 to 6.3], Standard Error of Mean 1.76 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported

4. Secondary Outcome: Percentage of Participants Achieving 50 Percent Reduction From Baseline PASI Score (PASI50 Response) at Weeks 2, 4, 6, 10 and 12
Description: PASI is an assessment of psoriasis lesion severity and affected body area combined into single score. The body was divided into 4 sections: head (h), trunk (t), upper (u) and lower (l) extremities. For each section, percent body surface area (A) involved was estimated: 0= No involvement to 6= 90-100 percent (%). Severity was estimated by clinical signs: erythema (E), induration (I), and desquamation (D); scale: 0= no symptoms to 4= very marked. Final PASI = 0.1(Eh + Ih + Dh)Ah + 0.3(Et + It + Dt)At + 0.2(Eu + Iu + Du)Au + 0.4(El + Il + Dl)Al where head: 0.1, upper extremities (arms): 0.2, trunk: 0.3, lower extremities (legs): 0.4 (corresponding to approximately 10%, 20%, 30%, and 40% of body surface area, respectively); total possible score range: 0= no disease to 72= maximal disease. Participants showing at least 50% reduction in PASI score relative to baseline PASI Score are reported.
Time Frame: Weeks 2, 4, 6, 10 and 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg
Number analyzed (Participants) | 24 | 24 | 24 | 25 | 25
percentage of participants
  Week 2 (n= 24, 24, 24, 25, 25) | 4.2 | 0 | 0 | 0 | 0
  Week 4 (n= 24, 24, 23, 24, 24) | 8.3 | 4.2 | 8.7 | 4.2 | 0
  Week 6 (n= 23, 23, 24, 24, 23) | 13.0 | 13.0 | 8.3 | 4.2 | 4.3
  Week 10 (n= 22, 22, 24, 24, 22) | 22.7 | 18.2 | 12.5 | 8.3 | 9.1
  Week 12 (n= 23, 21, 22, 19, 20) | 21.7 | 19.0 | 18.2 | 10.5 | 20.0
Statistical Analysis 1: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 20 mg; Week 12: CMH P-values are from a CMH Chi-Square test using a 2*2 contingency table of treatment and responder status controlling for visit; Test type: Superiority or Other; p = 0.827, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.027, 95% CI 2-sided [-0.265 to 0.211] — Risk difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 2: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 50 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.768, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.036, 95% CI 2-sided [-0.269 to 0.198] — Risk difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 3: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 80 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.338, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.112, 95% CI 2-sided [-0.330 to 0.106] — Risk difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 4: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 150 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.890, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.017, 95% CI 2-sided [-0.261 to 0.226] — Risk difference (namilumab - placebo) and corresponding 95% confidence interval were reported

5. Secondary Outcome: Percentage of Participants Achieving 90 Percent Reduction From Baseline PASI Score (PASI90 Response) at Weeks 2, 4, 6, 10 and 12
Description: PASI is an assessment of psoriasis lesion severity and affected body area combined into single score. The body was divided into 4 sections: head (h), trunk (t), upper (u) and lower (l) extremities. For each section, percent body surface area (A) involved was estimated: 0= No involvement to 6= 90-100 percent (%). Severity was estimated by clinical signs: erythema (E), induration (I), and desquamation (D); scale: 0= no symptoms to 4= very marked. Final PASI = 0.1(Eh + Ih + Dh)Ah + 0.3(Et + It + Dt)At + 0.2(Eu + Iu + Du)Au + 0.4(El + Il + Dl)Al where head: 0.1, upper extremities (arms): 0.2, trunk: 0.3, lower extremities (legs): 0.4 (corresponding to approximately 10%, 20%, 30%, and 40% of body surface area, respectively); total possible score range: 0= no disease to 72= maximal disease. Participants showing at least 90% reduction in PASI score relative to baseline PASI Score are reported.
Time Frame: Weeks 2, 4, 6, 10 and 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg
Number analyzed (Participants) | 24 | 24 | 24 | 25 | 25
percentage of participants
  Week 2 (n= 24, 24, 24, 25, 25) | 0 | 0 | 0 | 0 | 0
  Week 4 (n= 24, 24, 23, 24, 24) | 0 | 0 | 0 | 0 | 0
  Week 6 (n= 23, 23, 24, 24, 23) | 0 | 4.3 | 0 | 0 | 0
  Week 10 (n= 22, 22, 24, 24, 22) | 0 | 4.5 | 0 | 0 | 0
  Week 12 (n= 23, 21, 22, 19, 20) | 0 | 4.8 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 20 mg; Week 12:CMH P-values are from a CMH Chi-Square test using a 2*2 contingency table of treatment and responder status controlling for visit; Test type: Superiority or Other; p = 0.295, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.048, 95% CI 2-sided [-0.043 to 0.139] — Risk difference (namilumab - placebo) and corresponding 95% confidence interval were reported

6. Secondary Outcome: Percentage of Participants Achieving Greater Than or Equal to (>=) 2 Point Improvement From Baseline in Static Physicians Global Assessment (sPGA) Score at Weeks 2, 4, 6, 10 and 12
Description: sPGA for psoriasis is scored on a 6-point scale, reflecting a global consideration of the erythema, plaque elevation and skin scaling across all psoriatic lesions. sPGA of psoriasis scale ranges from 0 (clear) to 5 (very severe). Participants who had >=2 point improvement are reported.
Time Frame: Weeks 2, 4, 6, 10 and 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg
Number analyzed (Participants) | 24 | 24 | 24 | 25 | 25
percentage of participants
  Week 2 (n= 24, 24, 24, 25, 25) | 0 | 0 | 0 | 0 | 0
  Week 4 (n= 24, 24, 23, 24, 24) | 0 | 4.2 | 4.3 | 0 | 0
  Week 6 (n= 23, 23, 24, 24, 23) | 0 | 13.0 | 4.2 | 0 | 0
  Week 10 (n= 22, 22, 24, 24, 22) | 13.6 | 4.5 | 4.2 | 0 | 4.5
  Week 12 (n= 23, 21, 22, 19, 20) | 13.0 | 14.3 | 9.1 | 0 | 5.0
Statistical Analysis 1: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 20 mg; Week 12: CMH P-values are from a CMH Chi-Square test using a 2*2 contingency table of treatment and sPGA response category controlling for visit; Test type: Superiority or Other; p = 0.906, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.012, 95% CI 2-sided [-0.191 to 0.216] — Risk difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 2: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 50 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.677, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.040, 95% CI 2-sided [-0.222 to 0.143] — Risk difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 3: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 80 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.107, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.130, 95% CI 2-sided [-0.268 to 0.007] — Risk difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 4: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 150 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.371, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.080, 95% CI 2-sided [-0.248 to 0.087] — Risk difference (namilumab - placebo) and corresponding 95% confidence interval were reported

7. Secondary Outcome: Percentage of Participants Achieving a sPGA Response of Clear (0) or Almost Clear (1) at Weeks 2, 4, 6, 10 and 12
Description: sPGA for psoriasis is scored on a 6-point scale, reflecting a global consideration of the erythema, plaque elevation and skin scaling across all psoriatic lesions. sPGA of psoriasis scale ranges from 0 (clear) to 5 (very severe). 'Clear' and 'Almost clear' included all participants who had scored a 0 or 1.
Time Frame: Weeks 2, 4, 6, 10 and 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg
Number analyzed (Participants) | 24 | 24 | 24 | 25 | 25
percentage of participants
  Week 2 (n= 24, 24, 24, 25, 25) | 0 | 0 | 0 | 0 | 0
  Week 4 (n= 24, 24, 23, 24, 24) | 0 | 0 | 0 | 0 | 0
  Week 6 (n= 23, 23, 24, 24, 23) | 0 | 4.3 | 0 | 0 | 0
  Week 10 (n= 22, 22, 24, 24, 22) | 0 | 4.5 | 0 | 0 | 0
  Week 12 (n= 23, 21, 22, 19, 20) | 0 | 9.5 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 20 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.134, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.095, 95% CI 2-sided [-0.030 to 0.221] — Risk difference (namilumab - placebo) and corresponding 95% confidence interval were reported

8. Secondary Outcome: Change From Baseline in sPGA Score at Weeks 2, 4, 6, 10, and 12
Description: sPGA for psoriasis is scored on a 6-point scale, reflecting a global consideration of the erythema, plaque elevation and skin scaling across all psoriatic lesions. sPGA of psoriasis scale ranges from 0 (clear) to 5 (very severe).
Time Frame: Baseline, Weeks 2, 4, 6, 10, and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg
Number analyzed (Participants) | 24 | 24 | 24 | 25 | 25
units on a scale
  Baseline (n=24, 24, 24, 25, 25) | 3.5 (0.11) | 3.5 (0.11) | 3.6 (0.11) | 3.3 (0.11) | 3.6 (0.10)
  Change at Week 2 (n=24, 24, 24, 25, 25) | -0.1 (0.08) | -0.1 (0.08) | -0.2 (0.08) | -0.1 (0.08) | -0.1 (0.08)
  Change at Week 4 (n=24, 24, 23, 24, 24) | -0.1 (0.10) | -0.3 (0.10) | -0.2 (0.10) | -0.2 (0.10) | -0.3 (0.09)
  Change at Week 6 (n=23, 23, 24, 24, 23) | -0.3 (0.12) | -0.5 (0.12) | -0.3 (0.12) | -0.2 (0.12) | -0.2 (0.12)
  Change at Week 10 (n=22, 22, 24, 24, 22) | -0.4 (0.12) | -0.5 (0.12) | -0.4 (0.12) | -0.3 (0.12) | -0.5 (0.12)
  Change at Week 12 (n=23, 21, 22, 19, 20) | -0.4 (0.13) | -0.6 (0.13) | -0.6 (0.13) | -0.4 (0.13) | -0.5 (0.13)
Statistical Analysis 1: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 20 mg; Week 12: Post-baseline least squares means and p-values were from a MMRM model with main effect of study site, treatment, visit and interaction between visit and treatment as fixed effects, baseline value as a covariate with an unstructured covariance structure. Baseline least squares means and p-values were obtained using an analysis of variance (ANOVA) model with terms for treatment and study site; Test type: Superiority or Other; p = 0.258, MMRM; LS Mean Difference = -0.2, 95% CI 2-sided [-0.6 to 0.2], Standard Error of Mean 0.18 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 2: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 50 mg; Week 12: Post-baseline least squares means and p-values were from a MMRM model with main effect of study site, treatment, visit and interaction between visit and treatment as fixed effects, baseline value as a covariate with an unstructured covariance structure. Baseline least squares means and p-values were obtained using an ANOVA model with terms for treatment and study site; Test type: Superiority or Other; p = 0.365, MMRM; LS Mean Difference = -0.2, 95% CI 2-sided [-0.5 to 0.2], Standard Error of Mean 0.18 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 3: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 80 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.757, MMRM; LS Mean Difference = 0.1, 95% CI 2-sided [-0.3 to 0.4], Standard Error of Mean 0.18 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 4: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 150 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.825, MMRM; LS Mean Difference = 0.0, 95% CI 2-sided [-0.4 to 0.3], Standard Error of Mean 0.18 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported

9. Secondary Outcome: Change From Baseline in Affected Body Surface Area (BSA) at Weeks 2, 4, 6, 10, and 12
Description: Assessment of BSA with psoriasis was performed by means of the palm method, where the palm of the participant's hand represented 1% of BSA. The affected areas were then calculated by their size compared to the participant's palm.
Time Frame: Baseline, Weeks 2, 4, 6, 10, and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of total body surface area
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg
Number analyzed (Participants) | 24 | 24 | 24 | 25 | 25
percentage of total body surface area
  Baseline (n=24, 24, 24, 25, 25) | 23.09 (3.674) | 24.39 (3.485) | 26.16 (3.596) | 22.35 (3.497) | 21.84 (3.385)
  Change at Week 2 (n=24, 24, 24, 25, 25) | -0.59 (0.624) | -0.22 (0.591) | 0.21 (0.610) | -0.35 (0.594) | -0.26 (0.576)
  Change at Week 4 (n=24, 24, 23, 24, 24) | -0.86 (0.945) | -1.02 (0.923) | -0.24 (0.940) | -0.09 (0.923) | 0.25 (0.911)
  Change at Week 6 (n=23, 23, 24, 24, 23) | -1.78 (1.366) | -3.65 (1.351) | 0.43 (1.349) | 0.36 (1.340) | 0.12 (1.343)
  Change at Week 10 (n=22, 22, 24, 24, 22) | -3.24 (1.551) | -4.55 (1.542) | -0.63 (1.522) | 0.45 (1.513) | -0.51 (1.535)
  Change at Week 12 (n=23, 21, 22, 19, 20) | -3.29 (1.537) | -3.48 (1.553) | -1.70 (1.527) | 0.35 (1.559) | -0.51 (1.560)
Statistical Analysis 1: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 20 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.931, MMRM; LS Mean Difference = -0.19, 95% CI 2-sided [-4.48 to 4.10], Standard Error of Mean 2.163 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 2: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 50 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.459, MMRM; LS Mean Difference = 1.59, 95% CI 2-sided [-2.65 to 5.84], Standard Error of Mean 2.143 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 3: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 80 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.094, MMRM; LS Mean Difference = 3.65, 95% CI 2-sided [-0.63 to 7.93], Standard Error of Mean 2.161 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 4: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 150 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.203, MMRM; LS Mean Difference = 2.78, 95% CI 2-sided [-1.52 to 7.09], Standard Error of Mean 2.173 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported

10. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Itching Score at Weeks 2, 4, 6, 10, and 12
Description: Assessments were performed using a portable electronic device, which was kept and used by the participant throughout the duration of the study. Participants were asked to indicate their level of itching by marking a horizontal line with "No itch" at the left extreme and "Worst itch imaginable" at the right extreme (scale ranging from 0 - 10, but not shown on the line). Each assessment was intended to capture the severity of itching experienced during the previous 24 hours.
Time Frame: Baseline, Weeks 2, 4, 6, 10, and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg
Number analyzed (Participants) | 24 | 24 | 24 | 25 | 25
units on a scale
  Baseline (n=23, 23, 24, 25, 25) | 5.35 (0.633) | 5.28 (0.600) | 5.67 (0.610) | 6.08 (0.593) | 5.00 (0.575)
  Change at Week 2 (n=23, 23, 23, 25, 24) | -1.34 (0.441) | -1.15 (0.418) | -1.92 (0.427) | -1.42 (0.417) | -1.36 (0.402)
  Change at Week 4 (n=23, 23, 23, 23, 24) | -1.38 (0.501) | -1.46 (0.480) | -2.10 (0.486) | -1.66 (0.477) | -1.48 (0.462)
  Change at Week 6 (n=22, 22, 24, 22, 23) | -1.08 (0.502) | -1.54 (0.482) | -2.01 (0.485) | -1.57 (0.479) | -1.33 (0.464)
  Change at Week 10 (n=21, 21, 24, 22, 21) | -1.12 (0.515) | -1.47 (0.497) | -2.00 (0.496) | -1.51 (0.492) | -1.68 (0.481)
  Change at Week 12 (n=22, 20, 22, 17, 20) | -0.95 (0.523) | -1.49 (0.508) | -2.11 (0.504) | -1.54 (0.508) | -2.11 (0.494)
Statistical Analysis 1: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 20 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.448, MMRM; LS Mean Difference = -0.53, 95% CI 2-sided [-1.92 to 0.86], Standard Error of Mean 0.700 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 2: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 50 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.099, MMRM; LS Mean Difference = -1.15, 95% CI 2-sided [-2.53 to 0.22], Standard Error of Mean 0.692 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 3: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 80 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.396, MMRM; LS Mean Difference = -0.59, 95% CI 2-sided [-1.96 to 0.78], Standard Error of Mean 0.690 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 4: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 150 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.102, MMRM; LS Mean Difference = -1.15, 95% CI 2-sided [-2.54 to 0.23], Standard Error of Mean 0.697 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported

11. Secondary Outcome: Change From Baseline in VAS Joint Pain Score at Weeks 2, 4, 6, 10, and 12
Description: Assessments were performed using a portable electronic device, which was kept and used by the participant throughout the duration of the study. Participants were asked to indicate their severity of joint pain by marking a horizontal line with "No pain" at the left extreme and "Worst pain imaginable" at the right extreme (scale ranging from 0 - 10, but not shown on the line). Each assessment was intended to capture the severity of pain experienced during the previous 24 hours.
Time Frame: Baseline, Weeks 2, 4, 6, 10, and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg
Number analyzed (Participants) | 24 | 24 | 24 | 25 | 25
units on a scale
  Baseline (n=23, 23, 24, 25, 25) | 1.55 (0.618) | 3.45 (0.585) | 3.52 (0.595) | 3.14 (0.579) | 2.13 (0.560)
  Change at Week 2 (n=23, 23, 23, 25, 24) | -0.25 (0.334) | -0.89 (0.316) | -0.81 (0.323) | -0.68 (0.311) | -0.30 (0.301)
  Change at Week 4 (n=23, 23, 23, 23, 24) | -0.28 (0.378) | -1.06 (0.362) | -0.91 (0.366) | -0.89 (0.356) | -0.47 (0.346)
  Change at Week 6 (n=22, 21, 24, 22, 23) | -0.04 (0.405) | -0.84 (0.390) | -0.90 (0.391) | -0.63 (0.384) | -0.47 (0.374)
  Change at Week 10 (n=21, 21, 24, 22, 21) | -0.08 (0.417) | -0.60 (0.402) | -0.77 (0.401) | -0.56 (0.396) | -0.56 (0.387)
  Change at Week 12 (n=22, 20, 22, 17, 20) | 0.51 (0.458) | -0.54 (0.449) | -0.75 (0.444) | -0.47 (0.452) | -0.72 (0.436)
Statistical Analysis 1: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 20 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.099, MMRM; LS Mean Difference = -1.04, 95% CI 2-sided [-2.29 to -0.20], Standard Error of Mean 0.626 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 2: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 50 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.045, MMRM; LS Mean Difference = -1.26, 95% CI 2-sided [-2.49 to -0.03], Standard Error of Mean 0.619 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 3: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 80 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.118, MMRM; LS Mean Difference = -0.98, 95% CI 2-sided [-2.21 to 0.25], Standard Error of Mean 0.620 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 4: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 150 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.050, MMRM; LS Mean Difference = -1.22, 95% CI 2-sided [-2.44 to 0.00], Standard Error of Mean 0.616 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported

12. Secondary Outcome: Change From Baseline in VAS Morning Stiffness Score at Weeks 2, 4, 6, 10, and 12
Description: Assessments were performed using a portable electronic device, which was kept and used by the participant throughout the duration of the study. Participants were asked to indicate their level of morning stiffness by marking a horizontal line with "No stiffness" at the left extreme and "Very severe stiffness" at the right extreme (scale ranging from 0 - 10, but not shown on the line). Each assessment was intended to capture the severity of stiffness experienced by the participant since waking on that particular day.
Time Frame: Baseline, Weeks 2, 4, 6, 10, and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg
Number analyzed (Participants) | 23 | 24 | 24 | 25 | 25
units on a scale
  Baseline (n=23, 23, 24, 25, 25) | 1.73 (0.592) | 3.32 (0.561) | 3.33 (0.571) | 2.77 (0.555) | 2.32 (0.537)
  Change at Week 2 (n=23, 23, 23, 25, 24) | -0.22 (0.276) | -0.87 (0.266) | -0.91 (0.271) | -0.67 (0.259) | -0.32 (0.250)
  Change at Week 4 (n=23, 23, 23, 23, 24) | -0.31 (0.316) | -0.95 (0.307) | -0.97 (0.310) | -0.80 (0.300) | -0.26 (0.291)
  Change at Week 6 (n=22, 21, 24, 22, 23) | -0.27 (0.351) | -0.84 (0.343) | -0.97 (0.342) | -0.61 (0.335) | -0.21 (0.327)
  Change at Week 10 (n=21, 21, 24, 22, 21) | -0.38 (0.372) | -0.74 (0.364) | -0.94 (0.362) | -0.46 (0.356) | -0.24 (0.349)
  Change at Week 12 (n=22, 20, 22, 17, 20) | -0.16 (0.368) | -0.79 (0.363) | -1.02 (0.359) | -0.43 (0.361) | -0.24 (0.350)
Statistical Analysis 1: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 20 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.211, MMRM; LS Mean Difference = -0.63, 95% CI 2-sided [-1.63 to 0.36], Standard Error of Mean 0.503 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 2: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 50 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.087, MMRM; LS Mean Difference = -0.86, 95% CI 2-sided [-1.85 to 0.13], Standard Error of Mean 0.497 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 3: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 80 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.580, MMRM; LS Mean Difference = -0.27, 95% CI 2-sided [-1.26 to 0.71], Standard Error of Mean 0.494 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 4: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 150 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.873, MMRM; LS Mean Difference = -0.08, 95% CI 2-sided [-1.06 to 0.90], Standard Error of Mean 0.496 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported

13. Secondary Outcome: Change From Baseline in Duration of Morning Stiffness at Weeks 2, 4, 6, 10, and 12
Description: Assessments were performed using a portable electronic device, which was kept and used by the participant throughout the duration of the study. Duration of stiffness was elicited in response to a standard question included in the portable device.
Time Frame: Baseline, Weeks 2, 4, 6, 10, and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg
Number analyzed (Participants) | 13 | 17 | 17 | 18 | 18
minutes
  Baseline (n=13, 17, 17, 18, 18) | 6.6 (5.65) | 14.2 (4.49) | 18.2 (4.84) | 16.6 (4.58) | 12.4 (4.91)
  Change at Week 2 (n=13, 16, 17, 17, 17) | 1.2 (3.33) | -1.7 (2.67) | 0.1 (2.85) | -5.3 (2.73) | -0.2 (2.88)
  Change at Week 4 (n=13, 16, 16, 16, 17) | -0.9 (3.49) | -3.0 (2.80) | 2.4 (3.01) | -2.8 (2.88) | 1.0 (3.03)
  Change at Week 6 (n=13, 13, 17, 14, 16) | -0.6 (4.06) | -2.4 (3.39) | 4.1 (3.50) | -2.0 (3.44) | 1.8 (3.55)
  Change at Week 10 (n=11, 15, 17, 15, 13) | -0.9 (4.30) | -2.3 (3.58) | 5.2 (3.71) | -2.0 (3.64) | 1.3 (3.77)
  Change at Week 12 (n=13, 14, 16, 12, 12) | -1.4 (5.12) | -3.0 (4.35) | 6.5 (4.44) | -0.6 (4.42) | 3.0 (4.56)
Statistical Analysis 1: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 20 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.803, MMRM; LS Mean Difference = -1.7, 95% CI 2-sided [-15.2 to 11.8], Standard Error of Mean 6.70 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 2: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 50 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.248, MMRM; LS Mean Difference = 7.9, 95% CI 2-sided [-5.7 to 21.4], Standard Error of Mean 6.73 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 3: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 80 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.914, MMRM; LS Mean Difference = 0.7, 95% CI 2-sided [-12.7 to 14.2], Standard Error of Mean 6.67 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 4: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 150 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.523, MMRM; LS Mean Difference = 4.3, 95% CI 2-sided [-9.2 to 17.9], Standard Error of Mean 6.74 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported

14. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Week 12
Description: The DLQI is a 10-point rating scale for determining the impact of dermatological conditions on the participant's quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). Maximum total score is 30, where 0-1 represents "No effect at all on participant's life" and 21-30 "Extremely large effect on participant's life" - higher scores indicating poorer quality of life.
Time Frame: Baseline, Week 12
Population: FAS where baseline and Week 12 assessment were available. FAS included all randomized and treated participants who had at least one valid post-baseline assessment of PASI in the double-blind period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg
Number analyzed (Participants) | 21 | 21 | 22 | 19 | 19
units on a scale
  Baseline | 13.8 (1.95) | 12.2 (1.85) | 10.3 (1.83) | 13.9 (1.95) | 11.4 (1.89)
  Change at Week 12 | -0.7 (1.06) | -0.7 (1.01) | -1.9 (1.01) | -2.1 (1.06) | -2.8 (1.03)
Statistical Analysis 1: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 20 mg; Post-baseline least squares means and p-values were from an Analysis of covariance (ANCOVA) model with main effect of study site and treatment with baseline value as a covariate. Baseline least squares means and p-values were obtained using an ANOVA model with terms for treatment and study site; Test type: Superiority or Other; p = 0.978, ANCOVA; LS Mean Difference = 0.0, 95% CI 2-sided [-2.7 to 2.8], Standard Error of Mean 1.37 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 2: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 50 mg; Post-baseline least squares means and p-values were from an ANCOVA model with main effect of study site and treatment with baseline value as a covariate. Baseline least squares means and p-values were obtained using an ANOVA model with terms for treatment and study site; Test type: Superiority or Other; p = 0.389, ANCOVA; LS Mean Difference = -1.2, 95% CI 2-sided [-3.9 to 1.5], Standard Error of Mean 1.36 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 3: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 80 mg; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.316, ANCOVA; LS Mean Difference = -1.4, 95% CI 2-sided [-4.2 to 1.4], Standard Error of Mean 1.39 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 4: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 150 mg; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.142, ANCOVA; LS Mean Difference = -2.1, 95% CI 2-sided [-4.9 to 0.7], Standard Error of Mean 1.41 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported

15. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey (SF-36) at Week 12
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well-being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. These 8 aspects are summarized as physical and mental health summary scores. The score range for the physical and mental health scores is 0-100 (100=highest level of functioning).
Time Frame: Baseline, Week 12
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg
Number analyzed (Participants) | 20 | 20 | 22 | 19 | 18
units on a scale
  Physical Health Summary Score: Baseline | 52.9 (2.08) | 46.6 (1.97) | 49.0 (1.92) | 52.8 (2.04) | 50.7 (2.05)
  Physical Health Summary Score: Change at Week 12 | -0.5 (1.31) | -2.6 (1.24) | -0.8 (1.19) | 0.9 (1.28) | 0.4 (1.27)
  Mental Health Summary Score: Baseline | 43.7 (2.67) | 42.9 (2.53) | 42.8 (2.46) | 42.3 (2.61) | 46.0 (2.63)
  Mental Health Summary Score: Change at Week 12 | 0.9 (1.78) | 2.8 (1.69) | 1.5 (1.64) | 1.5 (1.75) | 1.6 (1.76)
Statistical Analysis 1: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 20 mg; Physical Health Summary Score: Post-baseline least squares means and p-values were from an ANCOVA model with main effect of study site and treatment with baseline value as a covariate. Baseline least squares means and p-values were obtained using an ANOVA model with terms for treatment and study site; Test type: Superiority or Other; p = 0.229, ANCOVA; LS Mean Difference = -2.1, 95% CI 2-sided [-5.6 to 1.4], Standard Error of Mean 1.73 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 2: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 50 mg; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.863, ANCOVA; LS Mean Difference = -0.3, 95% CI 2-sided [-3.6 to 3.0], Standard Error of Mean 1.65 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 3: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 80 mg; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.403, ANCOVA; LS Mean Difference = 1.4, 95% CI 2-sided [-1.9 to 4.7], Standard Error of Mean 1.67 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 4: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 150 mg; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.597, ANCOVA; LS Mean Difference = 0.9, 95% CI 2-sided [-2.5 to 4.4], Standard Error of Mean 1.74 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 5: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 20 mg; Mental Health Summary Score: Post-baseline least squares means and p-values were from an ANCOVA model with main effect of study site and treatment with baseline value as a covariate. Baseline least squares means and p-values were obtained using an ANOVA model with terms for treatment and study site; Test type: Superiority or Other; p = 0.416, ANCOVA; LS Mean Difference = 1.9, 95% CI 2-sided [-2.7 to 6.5], Standard Error of Mean 2.32 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 6: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 50 mg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.770, ANCOVA; LS Mean Difference = 0.7, 95% CI 2-sided [-3.8 to 5.1], Standard Error of Mean 2.24 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 7: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 80 mg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.798, ANCOVA; LS Mean Difference = 0.6, 95% CI 2-sided [-4.0 to 5.2], Standard Error of Mean 2.31 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 8: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 150 mg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.767, ANCOVA; LS Mean Difference = 0.7, 95% CI 2-sided [-4.1 to 5.5], Standard Error of Mean 2.40 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported

16. Secondary Outcome: Change From Baseline in EuroQoL Health Questionnaire (EQ-5D)- Index Score at Week 12
Description: EQ-5D-Index score is a generic, multidimensional, health-related, quality-of-life instrument. The profile allows participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The score ranges from -0.594 to 1.000. The higher score indicates a better health state perceived by the participant.
Time Frame: Baseline, Week 12
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg
Number analyzed (Participants) | 20 | 20 | 22 | 19 | 18
units on a scale
  Baseline | 0.86 (0.041) | 0.80 (0.038) | 0.84 (0.038) | 0.81 (0.040) | 0.87 (0.040)
  Change at Week 12 | -0.02 (0.033) | -0.04 (0.031) | -0.04 (0.030) | 0.01 (0.033) | 0.01 (0.033)
Statistical Analysis 1: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 20 mg; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.570, ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.11 to 0.06], Standard Error of Mean 0.043 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 2: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 50 mg; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.619, ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.10 to 0.06], Standard Error of Mean 0.042 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 3: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 80 mg; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.597, ANCOVA; LS Mean Difference = 0.02, 95% CI 2-sided [-0.06 to 0.11], Standard Error of Mean 0.043 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 4: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 150 mg; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.509, ANCOVA; LS Mean Difference = 0.03, 95% CI 2-sided [-0.06 to 0.12], Standard Error of Mean 0.044 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported

17. Secondary Outcome: Change From Baseline in EQ-5D-VAS Score at Week 12
Description: EQ-5D-VAS is a participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 mm ("Worst imaginable health state") to 100 mm ("Best imaginable health state"); higher scores indicate a better health state.
Time Frame: Baseline, Week 12
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: millimeter (mm)
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg
Number analyzed (Participants) | 16 | 17 | 20 | 17 | 16
millimeter (mm)
  Baseline | 76.8 (5.77) | 58.9 (5.13) | 67.2 (5.09) | 75.3 (5.42) | 74.3 (5.47)
  Change at Week 12 | 0.5 (3.99) | -0.5 (3.67) | 5.3 (3.51) | -1.4 (3.74) | -1.9 (3.77)
Statistical Analysis 1: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 20 mg; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.845, ANCOVA; LS Mean Difference = -1.0, 95% CI 2-sided [-11.7 to 9.6], Standard Error of Mean 5.32 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 2: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 50 mg; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.323, ANCOVA; LS Mean Difference = 4.8, 95% CI 2-sided [-4.8 to 14.4], Standard Error of Mean 4.80 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 3: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 80 mg; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.697, ANCOVA; LS Mean Difference = -1.9, 95% CI 2-sided [-11.7 to 7.8], Standard Error of Mean 4.89 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 4: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 150 mg; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.633, ANCOVA; LS Mean Difference = -2.4, 95% CI 2-sided [-12.6 to 7.7], Standard Error of Mean 5.10 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported

18. Secondary Outcome: Mean Change From Baseline in Nail Psoriasis Severity Index (NAPSI) Score at Weeks 2, 4, 6, 10, and 12
Description: The NAPSI quantifies severity of nail psoriasis by evaluating the presence or absence of psoriatic manifestations on the nail matrix (pitting, leukonychia, red spots on lunula, crumbling) and nail bed (onycholysis, splinter hemorrhages, subungual hyperkeratosis, oil drop [salmon patch dyschromia]). Each finger nail divided with imaginary lines into quadrants and scored for both nail matrix and nail bed psoriasis (range from 0 [absence of psoriasis] to 4 [presence of psoriasis in all 4 quadrants]). The total NAPSI score equals the sum of scores for all of the finger nails evaluated and ranges from 0 to 80. Higher scores = more severe psoriasis.
Time Frame: Baseline, Weeks 2, 4, 6, 10, and 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg
Number analyzed (Participants) | 24 | 24 | 24 | 25 | 25
units on a scale
  Baseline (n=24, 24, 24, 25, 25) | 14.5 (3.56) | 9.6 (3.37) | 15.6 (3.48) | 12.0 (3.39) | 12.5 (3.28)
  Change at Week 2 (n=24, 24, 24, 25, 25) | -0.8 (0.53) | 0.1 (0.50) | 0.8 (0.52) | 0.4 (0.50) | 0.1 (0.48)
  Change at Week 4 (n=24, 24, 23, 24, 24) | -1.5 (0.77) | 0.0 (0.75) | 1.4 (0.77) | 0.6 (0.75) | 0.1 (0.74)
  Change at Week 6 (n=23, 23, 24, 24, 23) | -1.5 (0.99) | -0.2 (0.98) | 1.2 (0.98) | 2.3 (0.97) | -0.7 (0.97)
  Change at Week 10 (n=22, 22, 24, 24, 21) | -2.4 (1.03) | -0.6 (1.02) | 0.8 (1.01) | 2.0 (1.00) | 0.6 (1.02)
  Change at Week 12 (n=23, 21, 22, 19, 20) | -1.5 (1.17) | -0.5 (1.18) | 0.9 (1.16) | 2.5 (1.17) | 1.0 (1.18)
Statistical Analysis 1: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 20 mg; Week 12: Post-baseline least squares means and p-values were from a MMRM model with main effect of study site,treatment,visit and interaction between visit and treatment as fixed effects,baseline value as a covariate with an unstructured covariance structure. Baseline least squares means and p-values were obtained using an ANOVA model with terms for treatment and study site; Test type: Superiority or Other; p = 0.537, MMRM; LS Mean Difference = 1.0, 95% CI 2-sided [-2.2 to 4.3], Standard Error of Mean 1.64 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 2: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 50 mg; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.142, MMRM; LS Mean Difference = 2.4, 95% CI 2-sided [-0.8 to 5.6], Standard Error of Mean 1.62 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 3: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 80 mg; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.015, MMRM; LS Mean Difference = 4.0, 95% CI 2-sided [0.8 to 7.3], Standard Error of Mean 1.63 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported
Statistical Analysis 4: Comparison: Double-Blind Period: Placebo vs Double-Blind Period: Namilumab 150 mg; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.121, MMRM; LS Mean Difference = 2.6, 95% CI 2-sided [-0.7 to 5.8], Standard Error of Mean 1.64 — LS mean difference (namilumab - placebo) and corresponding 95% confidence interval were reported

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug.
Description: At each clinic visit the investigator was required to document any occurrence of adverse events - including at specified visits abnormal laboratory, ECG and lung function test findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Follow-up Period: Placebo: Participants who received namilumab-matching placebo injections during the double-blind treatment were to be followed-up for 18 weeks after the last dose of study drug - whether administered in the double-blind period or open-label extension period.
- Follow-up Period: Namilumab 20 mg: Participants who received namilumab 20 mg injections during the double-blind treatment were to be followed-up for 18 weeks after the last dose of study drug - whether administered in the double-blind period or open-label extension period.
- Follow-up Period: Namilumab 50 mg: Participants who received namilumab 50 mg injections during the double-blind treatment were to be followed-up after the last dose of study drug - whether administered in the double-blind period or open-label extension period.
- Follow-up Period: Namilumab 80 mg: Participants who received namilumab 80 mg injections during the double-blind treatment were to be followed-up for 18 weeks after the last dose of study drug - whether administered in the double-blind period or open-label extension period.
- Follow-up: Namilumab 150 mg: Participants who received namilumab 150 mg injections during the double-blind treatment were to be followed-up for 18 weeks after the last dose of study drug - whether administered in the double-blind period or open-label extension period.
Arm/Group | Double-Blind Period: Placebo | Double-Blind Period: Namilumab 20 mg | Double-Blind Period: Namilumab 50 mg | Double-Blind Period: Namilumab 80 mg | Double-Blind Period: Namilumab 150 mg | Open-Label Period: Namilumab 80 mg | Open-Label Period: Namilumab 150 mg | Follow-up Period: Placebo | Follow-up Period: Namilumab 20 mg | Follow-up Period: Namilumab 50 mg | Follow-up Period: Namilumab 80 mg | Follow-up: Namilumab 150 mg
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/24 | 0/24 | 0/25 | 0/25 | 0/12 | 0/48 | 0/24 | 0/24 | 0/24 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 5/24 | 0/24 | 2/24 | 3/25 | 2/25 | 4/12 | 2/48 | 1/24 | 0/24 | 0/24 | 1/25 | 1/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Period: Placebo (N=24) | Double-Blind Period: Namilumab 20 mg (N=24) | Double-Blind Period: Namilumab 50 mg (N=24) | Double-Blind Period: Namilumab 80 mg (N=25) | Double-Blind Period: Namilumab 150 mg (N=25) | Open-Label Period: Namilumab 80 mg (N=12) | Open-Label Period: Namilumab 150 mg (N=48) | Follow-up Period: Placebo (N=24) | Follow-up Period: Namilumab 20 mg (N=24) | Follow-up Period: Namilumab 50 mg (N=24) | Follow-up Period: Namilumab 80 mg (N=25) | Follow-up: Namilumab 150 mg (N=25)
Hypertensive crisis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Period: Placebo (N=24) | Double-Blind Period: Namilumab 20 mg (N=24) | Double-Blind Period: Namilumab 50 mg (N=24) | Double-Blind Period: Namilumab 80 mg (N=25) | Double-Blind Period: Namilumab 150 mg (N=25) | Open-Label Period: Namilumab 80 mg (N=12) | Open-Label Period: Namilumab 150 mg (N=48) | Follow-up Period: Placebo (N=24) | Follow-up Period: Namilumab 20 mg (N=24) | Follow-up Period: Namilumab 50 mg (N=24) | Follow-up Period: Namilumab 80 mg (N=25) | Follow-up: Namilumab 150 mg (N=25)
Nasopharyngitis (Infections and infestations) | 3 | 0 | 1 | 3 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.